CLINICAL TRIAL: NCT03569293
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Upadacitinib in Adolescent and Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Evaluation of Upadacitinib in Adolescent and Adult Patients With Moderate to Severe Atopic Dermatitis (Eczema)
Acronym: Measure Up 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-045; 2022-502938-30-00 (Other: EU CT)
Expanded Access: NCT04159597 (Available)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2022-02-03 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Upadacitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo / Upadacitinib (Placebo Comparator): Participants will receive placebo orally once a day (QD) for 16 weeks in the double-blind treatment period. At Week 16 participants will be re-randomized to receive either upadacitinib 15 mg or upadacitinib 30 mg QD up to Week 260.
  Interventions: Drug: Placebo for Upadacitinib; Drug: Upadacitinib
- Upadacitinib 15 mg QD (Experimental): Participants will receive upadacitinib 15 mg orally once a day for up to 260 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 30 mg QD (Experimental): Participants will receive upadacitinib 30 mg orally once a day for up to 260 weeks.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo for Upadacitinib — Tablets taken orally once a day
  Arms: Placebo / Upadacitinib
Drug: Upadacitinib — Tablets taken orally once a day
  Other Names: ABT-494; RINVOQ™

SUMMARY:
The objective of this study is to assess the efficacy and safety of upadacitinib for the treatment of adolescent and adult participants with moderate to severe atopic dermatitis (AD) who are candidates for systemic therapy.

DETAILED DESCRIPTION:
This study includes a 35-day screening period, a 16-week double-blind period, a blinded extension period up to Week 260, and a 30-day follow-up visit.

Participants who meet eligibility criteria in the main study will be randomized in a 1:1:1 ratio to receive a daily oral dose of upadacitinib 30 mg or upadacitinib 15 mg or matching placebo. Upon completion of enrollment of 810 participants in the main study, a supplemental study will continue to enroll adolescents (adolescent sub-study) until a total of 180 adolescent participants are enrolled in the overall study (main study + adolescent sub-study).

Randomization for the main study will be stratified by baseline disease severity (validated Investigator Global Assessment scale for Atopic Dermatitis [vIGA-AD] score of moderate [3] versus severe [4]), by geographic region (United States [US]/Puerto Rico/Canada, Japan, China, and Other), and by age (adolescent [ages 12 to 17] versus adult [ages 18 to 75]). The separate randomization for the adolescent sub-study will be stratified by baseline disease severity (moderate [vIGA-AD 3] vs. severe [vIGA-AD 4]) and by geographic region (US/Puerto Rico/Canada and Other).

At Week 16 of the main study and the adolescent sub-study, participants in the placebo group will be re-randomized in a 1:1 ratio to receive daily oral doses of upadacitinib 30 mg or upadacitinib 15 mg in the blinded extension period. In the main study the re-randomization at Week 16 will be stratified by Week 16 50% improvement in Eczema Area and Severity Index [EASI 50] responder [yes/no], geographic region [US/Puerto Rico/Canada, China [Mainland], Japan, and other], and age group [adolescent/adult]. For the adolescent sub-study, the re-randomization will be stratified by EASI 50 responder (Yes/No) and by geographic region (US/Puerto Rico/Canada and Other).

Participants originally randomized to upadacitinib will continue upadacitinib in the extension period at the same dose.

Starting at the Week 4 visit, rescue treatment for AD may be provided at the discretion of the investigator if medically necessary.

The Primary Analysis for the main study will be conducted after all ongoing participants have completed Week 16. In addition, a Primary Analysis for the adolescent population (including the adolescent participants from the main study and the adolescent sub-study) will be conducted after all ongoing adolescent participants have completed Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of ≥ 40 kg at Baseline Visit for participants between ≥ 12 and < 18 years of age
* Chronic atopic dermatitis (AD) with onset of symptoms at least 3 years before Baseline Visit and subject meets Hanifin and Rajka criteria.
* Active moderate to severe AD defined by:

  * Eczema Area and Severity Index (EASI) score ≥ 16 at the Screening and Baseline Visits;
  * Validated Investigator's Global Assessment (vIGA) score ≥ 3 at the Screening and Baseline Visits;
  * ≥ 10% Body surface area (BSA) of AD involvement at the Screening and Baseline Visits;
  * Baseline weekly average of daily Worst Pruritus NRS ≥ 4.
* Candidate for systemic therapy or have recently required systemic therapy for AD
* Subject has applied a topical emollient (moisturizer) twice daily for at least 7 days before the Baseline Visit.
* Documented history of inadequate response to topical corticosteroids (TCS) or topical calcineurin inhibitor (TCI) or documented systemic treatment for AD within 6 months before Baseline Visit

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor
* Unable or unwilling to discontinue current atopic dermatitis treatments prior to the study
* Requirement of prohibited medications during the study
* Other active skin diseases or skin infections requiring systemic treatment or would interfere with appropriate assessment of atopic dermatitis lesions
* Female subject who is pregnant, breastfeeding, or considering pregnancy during the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2025-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (180):
- United States (58):
  - Alliance Dermatology and MOHs /ID# 200375, Phoenix, Arizona
  - Clear Dermatology & Aesthetics Center /ID# 201256, Scottsdale, Arizona
  - Bakersfield Derma & Skin Cance /ID# 200433, Bakersfield, California
  - First OC Dermatology /ID# 201910, Fountain Valley, California
  - California Allergy and Asthma Medical Group /ID# 200727, Los Angeles, California
  - Allergy & Asthma Associates of Southern California /ID# 200733, Mission Viejo, California
  - Dermatology Clinical Trials /ID# 205876, Newport Beach, California
  - UC Davis /ID# 203622, Sacramento, California
  - Synergy Dermatology /ID# 200842, San Francisco, California
  - San Luis Derm and Laser Clinic /ID# 200372, San Luis Obispo, California
  - Stanford University /ID# 200440, Stanford, California
  - Care Access Research - Walnut Creek /ID# 200940, Walnut Creek, California
  - Dermatology Physicians of Connecticut /ID# 200928, Shelton, Connecticut
  - Foxhall Research Center /ID# 213682, Washington D.C., District of Columbia
  - Duplicate_George Washington Univ Med /ID# 200364, Washington D.C., District of Columbia
  - Clearlyderm Dermatology /ID# 208371, Boca Raton, Florida
  - Skin Care Research, LLC /ID# 200811, Boca Raton, Florida
  - Olympian Clinical Research /ID# 202914, Clearwater, Florida
  - Multi-Speciality Research Associates /ID# 213254, Lake City, Florida
  - GSI Clinical Research, LLC /ID# 200849, Margate, Florida
  - Florida International Rsrch cr /ID# 218507, Miami, Florida
  - Tory P Sullivan, MD PA /ID# 200671, North Miami Beach, Florida
  - Leavitt Medical Associates of Florida /ID# 200880, Ormond Beach, Florida
  - Precision Clinical Research /ID# 209002, Sunrise, Florida
  - Integrated Clinical Research LLC /ID# 200900, West Palm Beach, Florida
  - Christie Clinic, LLC /ID# 200427, Champaign, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 201644, Chicago, Illinois
  - Dawes Fretzin, LLC /ID# 200366, Indianapolis, Indiana
  - The South Bend Clinic Center /ID# 200371, South Bend, Indiana
  - Clinical Trials Management, LLC - Covington /ID# 212658, Covington, Louisiana
  - Clinical Trials Management, LLC - Metairie /ID# 212659, Metairie, Louisiana
  - Northeast Dermatology /ID# 201338, Beverly, Massachusetts
  - Massachusetts General Hospital /ID# 200474, Boston, Massachusetts
  - Integrated Dermatology of Massachusetts, LLC /ID# 209468, Quincy, Massachusetts
  - Clin Res Inst of Michigan, LLC /ID# 208019, Chesterfield, Michigan
  - Henry Ford Medical Center /ID# 204191, Detroit, Michigan
  - Cleaver Dermatology /ID# 202825, Kirksville, Missouri
  - Advanced Dermatology of the Midlands /ID# 201689, Omaha, Nebraska
  - Clinical Research Consortium /ID# 200734, Las Vegas, Nevada
  - AllCutis Research Inc /ID# 200981, Portsmouth, New Hampshire
  - Forest Hills Dermatology Group /ID# 209244, Kew Gardens, New York
  - Icahn School of Medicine at Mount Sinai /ID# 200370, New York, New York
  - Montefiore Medical Center /ID# 200456, The Bronx, New York
  - J. Schwartz, MD, PLLC /ID# 202121, Troy, New York
  - Velocity clinical research /ID# 202653, Cleveland, Ohio
  - Lynn Health Science Institute (LHSI) /ID# 212676, Oklahoma City, Oklahoma
  - Newton Clinical Research /ID# 204169, Oklahoma City, Oklahoma
  - Oregon Medical Res Center PC /ID# 200428, Portland, Oregon
  - Oregon Health and Science University /ID# 200992, Portland, Oregon
  - Dermdox Dermatology Centers, PC /ID# 213782, Hazleton, Pennsylvania
  - Clinical Partners, LLC /ID# 200460, Johnston, Rhode Island
  - Coastal Clinical Research Center of the Carolinas /ID# 200402, Charleston, South Carolina
  - Arlington Research Center, Inc /ID# 200391, Arlington, Texas
  - Orion Clinical Research /ID# 204703, Austin, Texas
  - Modern Research Associates, PL /ID# 200705, Dallas, Texas
  - Menter Dermatology Res Inst /ID# 200390, Dallas, Texas
  - Center for Clinical Studies - Webster TX /ID# 203185, Webster, Texas
  - Dermatology Specialists of Spokane /ID# 202068, Spokane, Washington
- Argentina (3):
  - Framingham Centro Medico /ID# 202688, La Plata, Buenos Aires
  - Instituto de Neumonología y Dermatología /ID# 203444, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Psoriahue Med Interdisciplinar /ID# 202451, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
- Australia (5):
  - Woden Dermatology /ID# 205799, Phillip, Australian Capital Territory
  - Holdsworth House Medical Practice /ID# 211236, Darlinghurst, New South Wales
  - North Eastern Health Specialists /ID# 205802, Hectorville, South Australia
  - Skin Health Institute Inc /ID# 204791, Carlton, Victoria
  - Fremantle Dermatology /ID# 205305, Fremantle, Western Australia
- Bosnia and Herzegovina (4):
  - University Clinical Centre of the Republic of Srpska /ID# 202666, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 202667, Banja Luka, Republika Srpska
  - Clinical Center University of Sarajevo /ID# 202668, Sarajevo
  - Clinical Center University of Sarajevo /ID# 202669, Sarajevo
- Bulgaria (3):
  - UMHAT Alexandrovska EAD /ID# 201519, Sofiya, Sofia
  - UMHAT Dr Georgi Stranski EAD /ID# 201521, Pleven
  - UMHAT Professor Stoyan Kirkovich /ID# 201522, Stara Zagora
- Canada (15):
  - Kirk Barber Research, CA /ID# 200324, Calgary, Alberta
  - Dermatology Research Institute Inc. /ID# 200318, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 200311, Surrey, British Columbia
  - Enverus Medical Research /ID# 200307, Surrey, British Columbia
  - Wiseman Dermatology Research /ID# 200323, Winnipeg, Manitoba
  - Dr. Irina Turchin PC Inc. /ID# 200322, Fredericton, New Brunswick
  - Karma Clinical Trials /ID# 200316, St. John's, Newfoundland and Labrador
  - Hamilton Health Sciences - McMaster University Medical Centre /ID# 200313, Hamilton, Ontario
  - Dr. Wei Jing Loo Medicine Prof /ID# 206051, London, Ontario
  - Lynderm Research Inc. /ID# 200315, Markham, Ontario
  - Dermatology Ottawa Research Centre /ID# 200319, Ottawa, Ontario
  - K. Papp Clinical Research /ID# 200317, Waterloo, Ontario
  - Innovaderm Research Inc. /ID# 200320, Montreal, Quebec
  - Dr. David Gratton Dermat Inc. /ID# 200309, Montreal, Quebec
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 200326, Saint-Jérôme, Quebec
- China (10):
  - Peking University People's Hospital /ID# 202549, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 202612, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University /ID# 208597, Guangzhou, Guangdong
  - The Third Affiliated Hospital Of Sun Yat-Sen University /ID# 202548, Guangzhou, Guangdong
  - The First Hospital of China Medical University /ID# 202615, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 202554, Shanghai, Shanghai Municipality
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 202608, Hangzhou, Zhejiang
  - Beijing Friendship Hospital /ID# 202601, Beijing
  - Huashan Hospital of Fudan University /ID# 205760, Shanghai
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 208598, Wuhan
- Colombia (4):
  - Clinisalud del sur /ID# 218100, Medellín, Antioquia
  - Fundacion Hospital San Vicente de Paul - Rionegro /ID# 202043, Rionegro, Antioquia
  - Ctr Int de Reum del Caribe SAS /ID# 201620, Barranquilla, Atlántico
  - Fundacion Centro de Excelencia en Enfermedades Cronicas no Transmisibles - FUNCE /ID# 201905, Montería, Departamento de Córdoba
- Croatia (5):
  - Klinicki bolnicki centar Zagreb /ID# 201879, Zagreb, City of Zagreb
  - Klinika za dječje bolesti Zagreb /ID# 203151, Zagreb, City of Zagreb
  - Duplicate_Klinicki bolnicki centar Osijek /ID# 201523, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Rijeka /ID# 217423, Rijeka, Primorje-Gorski Kotar County
  - Klinicki bolnicki centar Split /ID# 201527, Split, Split-Dalmatia County
- Denmark (3):
  - Bispebjerg and Frederiksberg Hospital /ID# 200979, Copenhagen NV, Capital Region
  - Herlev and Gentofte Hospital /ID# 200736, Hellerup, Capital Region
  - Aarhus University Hospital /ID# 200737, Aarhus N, Central Jutland
- Estonia (3):
  - North Estonia Medical Centre /ID# 200951, Mustamäe, Harju
  - Confido Private Medical Clinic /ID# 200846, Tallinn, Harju
  - Tartu University Hospital /ID# 200847, Tartu, Tartu
- Finland (3):
  - Mehiläinen Neo /ID# 201116, Turku, Southwest Finland
  - Kuopio University Hospital /ID# 202449, Kuopio
  - Terveystalo Tampere /ID# 201117, Tampere
- France (8):
  - HCL - Hôpital Lyon Sud /ID# 201529, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU de Nantes, Hotel Dieu -HME /ID# 206377, Nantes, Pays de la Loire Region
  - Centre Hospitalier du Mans /ID# 205991, Le Mans, Sarthe
  - Hopital Saint Vincent de Paul /ID# 218253, Lille
  - Le Bateau BLanc /ID# 206833, Martigues
  - AP-HP - Hopital Necker /ID# 218364, Paris
  - Hôpital Charles-Nicolle /ID# 201525, Rouen
  - CHU Toulouse - Hopital Larrey /ID# 201528, Toulouse
- Germany (9):
  - Duplicate_Klinikum rechts der Isar - Technische Universitaet Muenchen /ID# 202087, Munich, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 202089, Frankfurt am Main, Hesse
  - Universitaetsklinikum Muenster /ID# 202085, Münster, North Rhine-Westphalia
  - CMS3 Company for Medical Study /ID# 205193, Selters, Rhineland-Palatinate
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 202255, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Bonn /ID# 202086, Bonn
  - TFS Trial Form Support GmbH /ID# 202083, Hamburg
  - Medizinische Hochschule Hannover /ID# 202091, Hanover
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz /ID# 205192, Mainz
- Italy (6):
  - Fondazione PTV Policlinico Tor Vergata /ID# 201136, Rome, Roma
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 200692, Ancona
  - A.O.U. di Bologna Policlinico S.Orsola-Malpighi /ID# 200746, Bologna
  - A.O.U. Policlinico G. Rodolico S.Marco- Presidio G.Rodolico /ID# 200741, Catania
  - Azienda Ospedaliera Universitaria Federico II /ID# 200750, Napoli
  - Azienda Ospedaliero Universitaria Pisana-Stabilimento di Santa Chiara /ID# 200695, Pisa
- Japan (11):
  - Aichi Medical University Hospital /ID# 202833, Nagakute-shi, Aichi-ken
  - Fukuoka University Hospital /ID# 201309, Fukuoka, Fukuoka
  - Kyushu Central Hospital of the Mutual Aid Association of Public School Teachers /ID# 202891, Fukuoka, Fukuoka
  - Gifu University Hospital /ID# 201760, Gifu, Gifu
  - Ogaki Municipal Hospital /ID# 203463, Ogaki-shi, Gifu
  - Takagi Dermatology Clinic /ID# 201238, Obihiro-shi, Hokkaido
  - Medical Cooperation Kojinkai Sapporo Skin Clinic /ID# 201239, Sapporo, Hokkaido
  - University Hospital Kyoto Prefectural University of Medicine /ID# 201876, Kyoto, Kyoto
  - Kume Clinic /ID# 201912, Sakai-shi, Osaka
  - NTT Medical Center Tokyo /ID# 201759, Shinagawa-ku, Tokyo
  - University of Yamanashi Hospital /ID# 204174, Chuo-shi, Yamanashi
- Malaysia (3):
  - Hospital Raja Permaisuri Bainun /ID# 204375, Ipoh, Perak
  - Queen Elizabeth Hospital /ID# 204379, Division Pantai Barat Utara, Sabah
  - Hospital Selayang /ID# 204378, Batu Caves, Selangor
- Clinical Trials NZ /ID# 205335, Hamilton, New Zealand
- Puerto Rico (3):
  - Cruz-Santana, Carolina, PR /ID# 201096, Carolina
  - Ponce Medical School Foundation /ID# 201821, Ponce
  - Clinical Research Puerto Rico /ID# 203309, San Juan
- Romania (2):
  - Spitalul Clinic Colentina /ID# 205860, Bucharest
  - Cabinet Medical de Dermatovenerologie Dr. Remus Orasan /ID# 205862, Cluj-Napoca
- Russia (5):
  - Chelyabinsk Regional Clinical Dermatovenerologic Dispensary /ID# 201996, Chelyabinsk, Chelyabinsk Oblast
  - Clinical Dermatovenerology Dispensary /ID# 203439, Krasnodar, Krasnodarskiy Kray
  - Saratov State Medical University n.a. V.I. Razumovskiy /ID# 201595, Saratov, Saratov Oblast
  - Ural Research Institute of dermatovenerology and immunopathology /ID# 201593, Yekaterinburg, Sverdlovsk Oblast
  - National Medical Research Center for Children's Health /ID# 203440, Moscow
- Switzerland (5):
  - Universitätsspital Basel /ID# 201599, Basel, Canton of Basel-City
  - Hôpitaux Universitaires Genève /ID# 201600, Geneva, Canton of Geneva
  - CHUV, Centre hospitalier universitaire vaudois /ID# 200910, Lausanne, Canton of Vaud
  - CHUV, Centre hospitalier universitaire vaudois /ID# 206505, Lausanne, Canton of Vaud
  - Inselspital, Universitätsspital Bern /ID# 201598, Bern
- Turkey (Türkiye) (4):
  - Erciyes University Medical Fac /ID# 204098, Melikgazi, Kayseri
  - Hacettepe University Faculty of Medicine /ID# 204099, Ankara
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty /ID# 204100, Istanbul
  - Gazi Universitesi Tip Fakultes /ID# 204176, Yenimahalle
- Ukraine (2):
  - Military Hospital of Military-Medical Clinical Center of Southern Region /ID# 201962, Zaporizhzhya, Zaporizhzhia Oblast
  - ME "Rivne Regional Dermatology and Venereology Dispensary" of RRC /ID# 210504, Rivne
- United Kingdom (5):
  - West Middlesex University Hospital /ID# 202273, Isleworth, London, City of
  - Barts Health NHS Trust /ID# 201043, London, London, City of
  - Guy's and St Thomas' NHS Foundation Trust /ID# 201192, London, London, City of
  - Chelsea and Westminster Hospital NHS Foundation Trust9 /ID# 201971, London
  - Northern Care Alliance NHS Group /ID# 201194, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Irvine AD, Prajapati VH, Guttman-Yassky E, Simpson EL, Papp KA, Blauvelt A, Chu CY, Hong HC, Gold LFS, de Bruin-Weller M, Bieber T, Kabashima K, Rosmarin D, Sancho C, Calimlim BM, Grada A, Yang Y, Wu X, Levy G, Raymundo EM, Teixeira HD, Silverberg JI. Efficacy and Safety of Upadacitinib in Patients With Moderate-to-Severe Atopic Dermatitis: Phase 3 Randomized Clinical Trial Results Through 140 Weeks. Am J Clin Dermatol. 2025 Nov;26(6):1003-1016. doi: 10.1007/s40257-025-00975-3. Epub 2025 Sep 3. PMID 40900410
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Simpson EL, Silverberg JI, Prajapati VH, Eyerich K, Katoh N, Boguniewicz M, Guttman-Yassky E, Song EJ, Lee WJ, Teixeira HD, Wu T, Sancho Sanchez C, Vigna N, Calimlim BM, de Bruin-Weller M. Rapid Itch Improvement and Skin Clearance with Upadacitinib Versus Placebo (Measure Up 1 and Measure Up 2) and Versus Dupilumab (Heads Up): Results from Three Phase 3 Clinical Trials in Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Aug;15(8):2061-2076. doi: 10.1007/s13555-025-01443-w. Epub 2025 Jun 2. PMID 40457140
- [Derived] Paller AS, Mendes-Bastos P, Siegfried E, Eichenfield LF, Soong W, Prajapati VH, Lio P, Simpson EL, Raymundo EM, Suravaram S, Hu X, Yang Y, Huang X, Calimlim BM, Platt AM, Su JC, Zheng M, Yamamoto-Hanada K, Teixeira HD, Irvine AD. Upadacitinib in Adolescents With Moderate to Severe Atopic Dermatitis: Analysis of 3 Phase 3 Randomized Clinical Trials Through 76 Weeks. JAMA Dermatol. 2024 Dec 1;160(12):1304-1313. doi: 10.1001/jamadermatol.2024.3696. PMID 39441580
- [Derived] Blauvelt A, Eyerich K, Irvine AD, de Bruin-Weller M, Kwatra SG, Gooderham M, Kim B, Calimlim BM, Lee WJ, Raymundo EM, Liu Y, Ofori S, Platt AM, Silverberg JI. More Time Spent with Clear Skin and No Itch with Upadacitinib versus Dupilumab for Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2621-2630. doi: 10.1007/s13555-024-01242-9. Epub 2024 Aug 7. PMID 39110139
- [Derived] Simpson EL, Prajapati VH, Leshem YA, Chovatiya R, de Bruin-Weller MS, Stander S, Pink AE, Calimlim BM, Lee WJ, Teixeira H, Ladizinski B, Hu X, Yang Y, Liu Y, Liu M, Grada A, Platt AM, Silverberg JI. Upadacitinib Rapidly Improves Patient-Reported Outcomes in Atopic Dermatitis: 16-Week Results from Phase 3 Clinical Trials (Measure Up 1 and 2). Dermatol Ther (Heidelb). 2024 May;14(5):1127-1144. doi: 10.1007/s13555-024-01157-5. Epub 2024 May 2. PMID 38696027
- [Derived] Silverberg JI, Gooderham MJ, Paller AS, Deleuran M, Bunick CG, Gold LFS, Hijnen D, Calimlim BM, Lee WJ, Teixeira HD, Hu X, Zhang S, Yang Y, Grada A, Platt AM, Thaci D. Early and Sustained Improvements in Symptoms and Quality of Life with Upadacitinib in Adults and Adolescents with Moderate-to-Severe Atopic Dermatitis: 52-Week Results from Two Phase III Randomized Clinical Trials (Measure Up 1 and Measure Up 2). Am J Clin Dermatol. 2024 May;25(3):485-496. doi: 10.1007/s40257-024-00853-4. Epub 2024 Mar 25. PMID 38528257
- [Derived] Thyssen JP, Thaci D, Bieber T, Gooderham M, de Bruin-Weller M, Soong W, Kabashima K, Barbarot S, Luna PC, Xu J, Hu X, Liu Y, Raymundo EM, Calimlim BM, Nduaka C, Gamelli A, Simpson EL. Upadacitinib for moderate-to-severe atopic dermatitis: Stratified analysis from three randomized phase 3 trials by key baseline characteristics. J Eur Acad Dermatol Venereol. 2023 Sep;37(9):1871-1880. doi: 10.1111/jdv.19232. Epub 2023 Jun 21. PMID 37247226
- [Derived] Paller AS, Ladizinski B, Mendes-Bastos P, Siegfried E, Soong W, Prajapati VH, Lio P, Thyssen JP, Simpson EL, Platt AM, Raymundo EM, Liu J, Calimlim BM, Huang X, Gu Y, Hu X, Yang Y, Su JC, Zheng M, Yamamoto-Hanada K, Teixeira HD, Irvine AD. Efficacy and Safety of Upadacitinib Treatment in Adolescents With Moderate-to-Severe Atopic Dermatitis: Analysis of the Measure Up 1, Measure Up 2, and AD Up Randomized Clinical Trials. JAMA Dermatol. 2023 May 1;159(5):526-535. doi: 10.1001/jamadermatol.2023.0391. PMID 37043227
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Mendes-Bastos P, Ladizinski B, Guttman-Yassky E, Jiang P, Liu J, Prajapati VH, Simpson EL, Vigna N, Teixeira HD, Barbarot S. Characterization of acne associated with upadacitinib treatment in patients with moderate-to-severe atopic dermatitis: A post hoc integrated analysis of 3 phase 3 randomized, double-blind, placebo-controlled trials. J Am Acad Dermatol. 2022 Oct;87(4):784-791. doi: 10.1016/j.jaad.2022.06.012. Epub 2022 Jun 15. PMID 35714786
- [Derived] Simpson EL, Papp KA, Blauvelt A, Chu CY, Hong HC, Katoh N, Calimlim BM, Thyssen JP, Chiou AS, Bissonnette R, Stein Gold LF, Wegzyn C, Hu X, Liu M, Liu J, Tenorio AR, Chu AD, Guttman-Yassky E. Efficacy and Safety of Upadacitinib in Patients With Moderate to Severe Atopic Dermatitis: Analysis of Follow-up Data From the Measure Up 1 and Measure Up 2 Randomized Clinical Trials. JAMA Dermatol. 2022 Apr 1;158(4):404-413. doi: 10.1001/jamadermatol.2022.0029. PMID 35262646
- [Derived] Guttman-Yassky E, Teixeira HD, Simpson EL, Papp KA, Pangan AL, Blauvelt A, Thaci D, Chu CY, Hong HC, Katoh N, Paller AS, Calimlim B, Gu Y, Hu X, Liu M, Yang Y, Liu J, Tenorio AR, Chu AD, Irvine AD. Once-daily upadacitinib versus placebo in adolescents and adults with moderate-to-severe atopic dermatitis (Measure Up 1 and Measure Up 2): results from two replicate double-blind, randomised controlled phase 3 trials. Lancet. 2021 Jun 5;397(10290):2151-2168. doi: 10.1016/S0140-6736(21)00588-2. Epub 2021 May 21. PMID 34023008
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 151 study sites in 24 countries across Europe, North and South America, Oceania, and the Asia-Pacific region.
  The study included a 16-week double-blind treatment period followed by an ongoing blinded extension period.
  The first 810 adults and adolescents enrolled constituted the Main Study; additional adolescents were enrolled in the Adolescent Substudy to ensure enrollment of a total of 180 adolescent participants overall.
  Results are reported up to Week 16.
Pre-assignment Details: Participants were randomized equally into 1 of 3 treatment groups, stratified by disease severity (validated Investigator Global Assessment Scale for Atopic Dermatitis [vIGA-AD] moderate [3] vs severe [4]), geographic region (US/Puerto Rico/Canada, Japan, China, and Other), and age (adolescent [ages 12 to 17] vs adult [ages 18 to 75]). Randomization for the adolescent substudy was stratified by disease severity (vIGA-AD 3 vs vIGA-AD 4) and geographic region (US/Puerto Rico/Canada vs Other).
Groups:
- Adults: Placebo: Participants ≥ 18 years old received placebo orally once a day (QD) for 16 weeks.
- Adults: Upadacitinib 15 mg QD: Participants ≥ 18 years old received upadacitinib 15 mg orally once a day for 16 weeks.
- Adults: Upadacitinib 30 mg QD: Participants ≥ 18 years old received upadacitinib 30 mg orally once a day for 16 weeks.
- Adolescents: Placebo: Adolescent participants (12 - 17 years old) received placebo orally once a day for 16 weeks.
- Adolescents: Upadacitinib 15 mg QD: Adolescent participants received upadacitinib 15 mg orally once a day for 16 weeks.
- Adolescents: Upadacitinib 30 mg QD: Adolescent participants received upadacitinib 30 mg orally once a day for 16 weeks.
Period: Overall Study
Arm/Group | Adults: Placebo | Adults: Upadacitinib 15 mg QD | Adults: Upadacitinib 30 mg QD | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Started (Randomized into study) | 241 | 239 | 243 | 61 | 64 | 64
Received Study Drug | 241 | 239 | 243 | 61 | 64 | 64
Completed (Completed Week 16) | 204 | 230 | 229 | 57 | 64 | 64
Not Completed | 37 | 9 | 14 | 4 | 0 | 0
Not completed — Adverse Event | 4 | 1 | 5 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 2 | 4 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 1 | 1 | 0 | 0
Not completed — Other | 8 | 2 | 1 | 1 | 0 | 0
Not completed — Ongoing at Time of Analysis | 8 | 1 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Adults: Placebo: Participants ≥ 18 years old received placebo orally once a day for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Adults: Placebo | Adults: Upadacitinib 15 mg QD | Adults: Upadacitinib 30 mg QD | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD | Total
Number analyzed (Participants) | 241 | 239 | 243 | 61 | 64 | 64 | 912
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (14.44) | 37.3 (14.80) | 36.7 (15.12) | 15.1 (1.70) | 15.5 (1.99) | 15.7 (1.63) | 32.7 (15.87)
Age, Customized [Count of Participants; unit: Participants]
  12 - 14 years | 0 | 0 | 0 | 23 | 22 | 15 | 60
  15 - 17 years | 0 | 0 | 0 | 38 | 42 | 49 | 129
  18 - < 40 years | 145 | 143 | 154 | 0 | 0 | 0 | 442
  40 - < 65 years | 85 | 83 | 74 | 0 | 0 | 0 | 242
  ≥ 65 years | 11 | 13 | 15 | 0 | 0 | 0 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 103 | 110 | 33 | 34 | 36 | 430
  Male | 127 | 136 | 133 | 28 | 30 | 28 | 482
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 27 | 34 | 10 | 13 | 19 | 133
  Not Hispanic or Latino | 211 | 212 | 209 | 51 | 51 | 45 | 779
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 2 | 0 | 0 | 3
  Asian | 62 | 57 | 61 | 10 | 12 | 10 | 212
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Black or African American | 16 | 20 | 7 | 6 | 6 | 0 | 55
  White | 157 | 153 | 163 | 41 | 45 | 50 | 609
  More than one race | 4 | 8 | 11 | 2 | 1 | 4 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Study Enrollment [Count of Participants; unit: Participants]
  Main Study | 241 | 239 | 243 | 40 | 42 | 42 | 847
  Adolescent Substudy | 0 | 0 | 0 | 21 | 22 | 22 | 65
Geographic Region [Count of Participants; unit: Participants]
  US/Puerto Rico/Canada | 108 | 107 | 108 | 31 | 33 | 33 | 420
  Japan | 13 | 14 | 14 | 1 | 1 | 2 | 45
  China | 13 | 13 | 15 | 1 | 1 | 2 | 45
  Other | 107 | 105 | 106 | 28 | 29 | 27 | 402
vIGA-AD [Count of Participants; unit: Participants] — The vIGA-AD was used to assess the severity of AD based on lesion appearance on the following scale:
  * 0-Clear: No inflammatory signs of AD;
  * 1-Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2-Mild: Slight but definite erythema, induration/papulation and/or lichenification. No oozing or crusting;
  * 3-Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4-Severe: Marked erythema, induration/papulation and/or lichenification, oozing or crusting may be present.
  Participants
    3 (Moderate) | 132 | 130 | 129 | 35 | 35 | 37 | 498
    4 (Severe) | 109 | 109 | 114 | 26 | 29 | 27 | 414
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  score on a scale | 28.39 (12.082) | 30.34 (12.651) | 29.06 (11.270) | 29.65 (14.054) | 30.70 (12.816) | 27.77 (10.625) | 29.28 (12.125)
Disease Duration since Diagnosis [Mean (Standard Deviation); unit: years] | 22.704 (15.9393) | 22.010 (16.6733) | 21.655 (15.0471) | 11.391 (5.0989) | 12.027 (4.5017) | 12.443 (4.4464) | 20.017 (14.8779)

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Percentage of Participants Achieving at Least a 75% Reduction in Eczema Area and Severity Index Score (EASI 75) From Baseline at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Time Frame: Baseline and Week 16
Population: The intent-to-treat population for the main study (ITT_M) includes all participants who were randomized in the main study (adults and adolescents). Non-responder imputation incorporating multiple imputation to handle missing data due to coronavirus disease 2019 pandemic (COVID-19) (NRI-C) was used.
  The pre-specified primary analysis included participants enrolled in the main study only; Efficacy analyses of adolescent participants were conducted separately and are reported below.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received placebo orally once a day for 16 weeks.
- Upadacitinib 15 mg QD: Participants received upadacitinib 15 mg orally once daily for 16 weeks.
- Upadacitinib 30 mg QD: Participants received upadacitinib 30 mg orally once daily for 16 weeks.
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 281 | 281 | 285
percentage of participants | 16.3 [12.0 to 20.7] | 69.6 [64.2 to 75.0] | 79.7 [75.0 to 84.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 30 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 63.4, 95% CI 2-sided [57.1 to 69.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 15 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 53.3, 95% CI 2-sided [46.4 to 60.2] — Response Rate Difference = Upadacitinib - Placebo

2. Primary Outcome: Main Study: Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) of 0 or 1 With a Reduction From Baseline of ≥ 2 Points at Week 16
Description: The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No inflammatory signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 281 | 281 | 285
percentage of participants | 8.4 [5.2 to 11.7] | 48.1 [42.3 to 54.0] | 62.0 [56.4 to 67.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 53.6, 95% CI 2-sided [47.2 to 60.0] — Response rate difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 39.8, 95% CI 2-sided [33.2 to 46.4] — Response rate difference = Upadacitinib - Placebo

3. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus Numerical Rating Scale (NRS) at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with Worst Pruritus NRS (weekly average) ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 272 | 274 | 280
percentage of participants | 11.8 [7.9 to 15.6] | 52.2 [46.3 to 58.1] | 60.0 [54.3 to 65.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 48.2, 95% CI 2-sided [41.3 to 55.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 40.5, 95% CI 2-sided [33.5 to 47.5] — Response Rate Difference = Upadacitinib - Placebo

4. Secondary Outcome: Main Study: Percentage of Participants Achieving a 90% Reduction From Baseline in EASI Score (EASI 90) at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 281 | 281 | 285
percentage of participants | 8.1 [4.9 to 11.3] | 53.1 [47.2 to 58.9] | 65.8 [60.2 to 71.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 57.8, 95% CI 2-sided [51.5 to 64.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 45.1, 95% CI 2-sided [38.6 to 51.7] — Response Rate Difference = Upadacitinib - Placebo

5. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 4
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 272 | 274 | 280
percentage of participants | 4.4 [2.0 to 6.9] | 51.5 [45.5 to 57.4] | 66.8 [61.3 to 72.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 62.3, 95% CI 2-sided [56.3 to 68.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 47.1, 95% CI 2-sided [40.7 to 53.4] — Response Rate Difference = Upadacitinib - Placebo

6. Secondary Outcome: Main Study: Percentage of Participants Achieving an EASI 75 Response at Week 2
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 75 response is defined as at least a 75% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 281 | 281 | 285
percentage of participants | 3.6 [1.4 to 5.7] | 38.1 [32.4 to 43.8] | 47.4 [41.6 to 53.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 43.9, 95% CI 2-sided [37.7 to 50.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 34.5, 95% CI 2-sided [28.6 to 40.5] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 1
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 272 | 274 | 280
percentage of participants | 0.4 [0.0 to 1.1] | 15.0 [10.7 to 19.2] | 19.6 [15.0 to 24.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 19.2, 95% CI 2-sided [14.6 to 23.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 14.6, 95% CI 2-sided [10.3 to 18.8] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 2
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
  The percentage of participants who had a 4-point or greater improvement from Baseline in Worst Pruritus NRS score at Day 2 was pre-specified as a ranked secondary endpoint for participants in the upadacitinib 30 mg group versus placebo group only.
Time Frame: Baseline and Day 2
Population: Intent-to-treat population for the main study with Worst Pruritus NRS (daily score) ≥ 4 at Baseline; Non-responder imputation with no special data handling for missing data due to COVID-19 (NRI-NC) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 270 | 275 | 279
percentage of participants | 3.7 [1.5 to 6.0] | 10.5 [6.9 to 14.2] | 11.8 [8.0 to 15.6]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 8.1, 95% CI 2-sided [3.8 to 12.5] — Response Rate Difference = Upadacitinib - Placebo

9. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 3
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
  The percentage of participants who had a 4-point or greater improvement in Worst Pruritus NRS score from Baseline at Day 3 was pre-specified as a ranked secondary endpoint for participants in the upadacitinib 15 mg group versus placebo group only.
Time Frame: Baseline and Day 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 270 | 275 | 279
percentage of participants | 3.3 [1.2 to 5.5] | 16.4 [12.0 to 20.7] | 21.1 [16.4 to 25.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 13.0, 95% CI 2-sided [8.1 to 17.8] — Response Rate Difference = Upadacitinib - Placebo

10. Secondary Outcome: Main Study: Percentage of Participants Experiencing a Flare During the Double-blind Treatment Period
Description: A flare, characterized as a clinically meaningful worsening in EASI, is defined as an increase in EASI score of ≥ 6.6 points from Baseline during the double-blind treatment period and prior to use of any rescue medication. Flare was assessed in participants with an EASI score of 65.4 or less at Baseline.
Time Frame: From first dose of study drug to Week 16
Population: Intent-to-treat population for the main study with an EASI score ≤ 65.4 at Baseline and at least one EASI post-baseline assessment prior to use of rescue medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 274 | 279 | 285
percentage of participants | 25.2 [20.0 to 30.3] | 1.1 [0.0 to 2.3] | 0.0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = -25.2, 95% CI 2-sided [-30.3 to -20.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = -24.1, 95% CI 2-sided [-29.3 to -18.9] — Response Rate Difference = Upadacitinib - Placebo

11. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 12 Points From Baseline in Atopic Dermatitis Impact Scale (ADerm-IS) Sleep Domain Score at Week 16
Description: The ADerm-IS is a 10-item patient reported outcome (PRO) questionnaire designed to assess a variety of impacts that participants experience from their AD.
  The ADerm-IS sleep domain consists of 3 questions designed to assess the impact of AD on sleep on a daily basis over a 24-hour recall period. The items include difficulty falling asleep, impact on sleep, and waking at night. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The ADerm-IS sleep domain score is the sum of the 3 item scores and ranges from 0 (no impact) to 30 (worst impact). The ADerm-IS sleep domain was analyzed based on weekly rolling averages of daily scores.
  The minimal clinically important difference for ADerm-IS sleep domain score is 12.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with ADerm-IS Sleep Domain score ≥ 12 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 220 | 218 | 218
percentage of participants | 13.2 [8.7 to 17.7] | 55.0 [48.4 to 61.6] | 66.1 [59.8 to 72.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 52.9, 95% CI 2-sided [45.2 to 60.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 41.8, 95% CI 2-sided [33.9 to 49.7] — Response Rate Difference = Upadacitinib - Placebo

12. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Atopic Dermatitis Symptom Scale (ADerm-SS) Skin Pain Score at Week 16
Description: The ADerm-SS is an 11-item PRO questionnaire designed to assess signs and symptoms that patients may experience due to AD using a 24-hour recall period. For the skin pain item participants were asked on a daily basis to indicate how bad their worst skin pain due to AD was in the past 24 hours on an NRS from 0 (no pain) to 10 (worst imaginable pain). The ADerm-SS skin pain score was analyzed using weekly rolling averages of daily scores. The minimal clinically important difference for ADerm-SS skin pain score is 4.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with ADerm-SS Skin Pain Score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 233 | 237 | 249
percentage of participants | 15.0 [10.4 to 19.6] | 53.6 [47.2 to 59.9] | 63.5 [57.5 to 69.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 48.6, 95% CI 2-sided [41.0 to 56.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 38.7, 95% CI 2-sided [30.9 to 46.5] — Response Rate Difference = Upadacitinib - Placebo

13. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 28 Points From Baseline in ADerm-SS 7-Item Total Symptom Score (TSS-7) at Week 16
Description: The ADerm-SS is an 11-item questionnaire designed to assess signs and symptoms that participants may experience due to AD using a 24-hour recall period. The 7-item total symptom score includes 7 symptoms (items 1-7 of the ADerm-SS), each assessed on a NRS from 0 (no symptom) to 10 (worst imaginable). The 7 symptoms included in the score are itch while asleep, itch while awake, skin pain (each assessed daily), skin cracking, skin cracking pain, dry skin, and skin flaking (assessed weekly). The TSS-7 score ranges from 0 to 70, with higher scores indicating worsening symptoms. The minimal clinically important difference for ADerm-SS TSS-7 is 28.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with ADerm-SS TSS-7 ≥ 28 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 226 | 233 | 246
percentage of participants | 15.0 [10.4 to 19.7] | 53.6 [47.2 to 60.1] | 67.9 [62.1 to 73.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 52.9, 95% CI 2-sided [45.4 to 60.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 38.3, 95% CI 2-sided [30.4 to 46.2] — Response Rate Difference = Upadacitinib - Placebo

14. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 11 Points From Baseline in ADerm-IS Emotional State Domain Score at Week 16
Description: The ADerm-IS is a 10-item PRO questionnaire designed to assess a variety of impacts that participants experience from their AD.
  ADerm-IS emotional state sums three items [Items 8-10] measuring self-consciousness, embarrassment, and sadness with a 7-day recall. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The emotional state domain score ranges from 0 to 30, where higher scores represent worst impact.
  The minimal clinically important difference for ADerm-IS emotional state domain score is 11.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with ADerm-IS Emotional State domain score ≥ 11 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 212 | 227 | 226
percentage of participants | 19.8 [14.4 to 25.2] | 62.6 [56.3 to 68.9] | 72.6 [66.7 to 78.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 52.5, 95% CI 2-sided [44.7 to 60.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 42.7, 95% CI 2-sided [34.4 to 50.9] — Response Rate Difference = Upadacitinib - Placebo

15. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 14 Points From Baseline in in ADerm-IS Daily Activities Domain Score at Week 16
Description: The ADerm-IS is a 10-item PRO questionnaire designed to assess a variety of impacts that participants experience from their AD.
  ADerm-IS daily activities sums four items measuring limitations of household, physical, and social activities, and difficulty concentrating with a 7-day recall. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The daily activities domain score ranges from 0 to 40, where higher scores represent worst impact.
  The minimal clinically important difference for the ADerm-IS daily activities domain score is 14.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with ADerm-IS Daily Activities Domain Score ≥ 14 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 197 | 203 | 205
percentage of participants | 20.3 [14.7 to 25.9] | 65.0 [58.5 to 71.6] | 73.2 [67.1 to 79.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 53.1, 95% CI 2-sided [44.9 to 61.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 44.7, 95% CI 2-sided [36.2 to 53.2] — Response Rate Difference = Upadacitinib - Placebo

16. Secondary Outcome: Main Study: Percentage of Participants Achieving a 100% Reduction From Baseline in EASI Score (EASI 100) at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 281 | 281 | 285
percentage of participants | 1.8 [0.2 to 3.3] | 16.7 [12.4 to 21.1] | 27.0 [21.9 to 32.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 25.3, 95% CI 2-sided [20.0 to 30.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 15.0, 95% CI 2-sided [10.4 to 19.6] — Response Rate Difference = Upadacitinib - Placebo

17. Secondary Outcome: Main Study: Percent Change From Baseline in Worst Pruritus NRS at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores. A negative change from Baseline indicates improvement.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with non-missing Baseline and Week 16 values; missing data were handled using a mixed-effect model with repeated measurements (MMRM) including observed measurements at all visits, except that measurements after any rescue medication were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 123 | 225 | 236
percent change | -26.06 [-36.66 to -15.46] | -62.79 [-71.60 to -53.99] | -72.04 [-80.69 to -63.39]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 30 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, Baseline vIGA-AD category and age in the model; Least Squares (LS) Mean Difference = -45.98, 95% CI 2-sided [-58.82 to -33.15], Standard Error of Mean 6.549 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 15 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for EU/EMA regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -36.74, 95% CI 2-sided [-49.66 to -23.81] — Difference = Upadacitinib - Placebo

18. Secondary Outcome: Main Study: Percent Change From Baseline in EASI Score at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1)] moderate [2], or severe [3]) for Redness (erythema, inflammation), Thickness (induration, papulation, swelling - acute eczema), Scratching (excoriation), and Lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 128 | 244 | 259
percent change | -40.71 [-45.18 to -36.23] | -80.24 [-83.99 to -76.49] | -87.74 [-91.42 to -84.06]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 30 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for EU/EMA regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -47.03, 95% CI 2-sided [-52.37 to -41.70], Standard Error of Mean 2.716 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -39.53, 95% CI 2-sided [-44.91 to -34.15], Standard Error of Mean 2.738 — Difference = Upadacitinib - Placebo

19. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Patient Oriented Eczema Measure (POEM) Total Score at Week 16
Description: The POEM is a 7-item, validated questionnaire used to assess disease symptoms in both children and adults. Participants respond to 7 questions, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency of occurrence during the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores are added to provide a total score ranging from 0 (clear) to 28 (very severe atopic eczema). A change in POEM score of 3.4 points is considered the minimal clinically important difference.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with POEM score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 276 | 278 | 280
percentage of participants | 22.8 [17.8 to 27.8] | 75.0 [69.9 to 80.1] | 81.4 [76.9 to 86.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 58.6, 95% CI 2-sided [51.9 to 65.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 52.3, 95% CI 2-sided [45.2 to 59.4] — Response Rate Difference = Upadacitinib - Placebo

20. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL.
  the DLQI was administered to participants who were ≥ 16 (16 to 75) years old at the time of the Screening visit.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study who were ≥ 16 years old at Screening with DLQI score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 250 | 254 | 256
percentage of participants | 29.0 [23.3 to 34.7] | 75.4 [70.1 to 80.8] | 82.0 [77.3 to 86.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 53.2, 95% CI 2-sided [45.9 to 60.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 46.7, 95% CI 2-sided [39.0 to 54.4] — Response Rate Difference = Upadacitinib - Placebo

21. Secondary Outcome: Main Study: Percent Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score at Week 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 125 | 239 | 253
percent change | -32.68 [-37.26 to -28.11] | -65.71 [-69.20 to -62.23] | -73.07 [-76.47 to -69.68]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -40.39, 95% CI 2-sided [-45.75 to -35.03], Standard Error of Mean 2.732 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -33.03, 95% CI 2-sided [-38.44 to -27.61], Standard Error of Mean 2.758 — Difference = Upadacitinib - Placebo

22. Secondary Outcome: Main Study: Percentage of Participants Achieving a Hospital Anxiety and Depression Scale-Anxiety (HADS-A) Score and Hospital Anxiety and Depression Scale-Depression (HADS-D) Score of < 8 at Week 16
Description: The HADS is a 14-item questionnaire, with seven items related to anxiety (HADS-A) and seven items related to depression (HADS-D). Each item is scored from 0 to 3; scores for each subscale range from 0 to 21, with higher scores indicating more distress. For each domain, scores 7 or lower are considered normal, 8 to 10 are borderline, and 11 or higher indicate clinical anxiety or depression.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with HADS-A ≥ 8 or HADS-D ≥ 8 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 126 | 145 | 144
percentage of participants | 14.3 [8.2 to 20.4] | 45.5 [37.4 to 53.6] | 49.2 [41.0 to 57.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 34.9, 95% CI 2-sided [24.8 to 45.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 31.5, 95% CI 2-sided [21.4 to 41.6] — Response Rate Difference = Upadacitinib - Placebo

23. Secondary Outcome: Main Study: Percentage of Participants Achieving a DLQI Score of 0 or 1 at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL. A score of 0 or 1 means that the disease has no effect at all.
  the DLQI was administered to participants who were ≥ 16 (16 to 75) years old at the time of the Screening visit.
Time Frame: Week 16
Population: Intent-to-treat population for the main study who were ≥ 16 years old at Screening with DLQI score ≥ 1 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 252 | 258 | 261
percentage of participants | 4.4 [1.9 to 7.0] | 30.3 [24.7 to 35.9] | 41.5 [35.5 to 47.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 37.3, 95% CI 2-sided [30.8 to 43.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 25.9, 95% CI 2-sided [19.7 to 32.1] — Response Rate Difference = Upadacitinib - Placebo

24. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 75 Response at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: The ITT population for adolescents (ITT_A) consists of all adolescent participants who are randomized in the main study or the adolescent sub-study. Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adolescents: Placebo: Adolescent participants received placebo orally once a day for 16 weeks.
- Adolescents: Upadacitinib 15 mg QD: Adolescent participants received upadacitinib 15 mg orally once daily for 16 weeks.
- Adolescents: Upadacitinib 30 mg QD: Adolescent participants received upadacitinib 30 mg orally once daily for 16 weeks.
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 61 | 64 | 64
percentage of participants | 11.5 [3.5 to 19.5] | 73.4 [62.6 to 84.3] | 78.1 [68.0 to 88.3]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 66.6, 95% CI 2-sided [53.8 to 79.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 62.0, 95% CI 2-sided [48.6 to 75.4] — Response Rate Difference = Upadacitinib - Placebo

25. Secondary Outcome: Adolescents: Percentage of Participants Achieving a vIGA-AD of 0 or 1 With a Reduction From Baseline of ≥ 2 Points at Week 16
Description: The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, possible oozing or crusting;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; possible oozing or crusting.
Time Frame: Baseline and Week 16
Population: The ITT population for adolescents; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 61 | 64 | 64
percentage of participants | 6.6 [0.3 to 12.8] | 45.3 [33.1 to 57.5] | 64.1 [52.3 to 75.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 57.4, 95% CI 2-sided [44.6 to 70.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 39.1, 95% CI 2-sided [25.6 to 52.6] — Response Rate Difference = Upadacitinib - Placebo

26. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Worst pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with Worst Pruritus NRS (weekly average) ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 62 | 62
percentage of participants | 10.0 [2.4 to 17.6] | 48.4 [35.9 to 60.8] | 56.5 [44.1 to 68.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 46.6, 95% CI 2-sided [32.6 to 60.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 38.7, 95% CI 2-sided [24.3 to 53.1] — Response Rate Difference = Upadacitinib - Placebo

27. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 90 Response at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 90 response is defined as at least a 90% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 61 | 64 | 64
percentage of participants | 3.3 [0.0 to 7.7] | 46.9 [34.6 to 59.1] | 67.2 [55.7 to 78.7]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 63.9, 95% CI 2-sided [51.8 to 75.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 43.8, 95% CI 2-sided [30.9 to 56.7] — Response Rate Difference = Upadacitinib - Placebo

28. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 4
Description: as for outcome 26
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 4
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 62 | 62
percentage of participants | 3.3 [0.0 to 7.9] | 48.4 [35.9 to 60.8] | 58.1 [45.8 to 70.3]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 54.7, 95% CI 2-sided [41.7 to 67.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 45.2, 95% CI 2-sided [32.0 to 58.3] — Response Rate Difference = Upadacitinib - Placebo

29. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 75 Response at Week 2
Description: as for outcome 6
Time Frame: Baseline and Week 2
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 61 | 64 | 64
percentage of participants | 3.3 [0.0 to 7.7] | 39.1 [27.1 to 51.0] | 50.4 [38.0 to 62.7]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 47.1, 95% CI 2-sided [34.0 to 60.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 35.9, 95% CI 2-sided [23.2 to 48.6] — Response Rate Difference = Upadacitinib - Placebo

30. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 1
Description: as for outcome 26
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 1
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 62 | 62
percentage of participants | 0.0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 9.7 [2.3 to 17.0] | 21.0 [10.8 to 31.1]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 21.0, 95% CI 2-sided [11.0 to 31.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 9.4, 95% CI 2-sided [2.5 to 16.4] — Response Rate Difference = Upadacitinib - Placebo

31. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 2
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Day 2
Population: Intent-to-treat population for adolescents with Worst Pruritus NRS (daily score) ≥ 4 at Baseline; Non-responder imputation with no special data handling for missing data due to COVID-19 was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 60 | 63
percentage of participants | 1.7 [0.0 to 5.0] | 8.3 [1.3 to 15.3] | 12.7 [4.5 to 20.9]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 11.0, 95% CI 2-sided [2.1 to 19.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.086, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 6.5, 95% CI 2-sided [-0.9 to 13.9] — Response Rate Difference = Upadacitinib - Placebo

32. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 3
Description: as for outcome 31
Time Frame: Baseline and Day 3
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 60 | 63
percentage of participants | 5.1 [0.0 to 10.7] | 16.7 [7.2 to 26.1] | 15.9 [6.8 to 24.9]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p = 0.045, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 10.8, 95% CI 2-sided [0.2 to 21.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.040, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 11.0, 95% CI 2-sided [0.5 to 21.5] — Response Rate Difference = Upadacitinib - Placebo

33. Secondary Outcome: Adolescents: Percentage of Participants Experiencing a Flare During the Double-blind Treatment Period
Description: A flare, characterized as a clinically meaningful worsening in EASI, is defined as an increase in EASI score of ≥ 6.6 points from Baseline during the double-blind treatment period and prior to use of any rescue medication. Flares were assessed in participants with an EASI score of 65.4 or less at Baseline.
Time Frame: From first dose of study drug to Week 16
Population: Intent-to-treat population for adolescents with an EASI score ≤ 65.4 at Baseline and at least one EASI post-baseline assessment prior to use of rescue medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 63 | 64
percentage of participants | 22.0 [11.5 to 32.6] | 0.0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 0.0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = -22.1, 95% CI 2-sided [-32.6 to -11.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = -22.1, 95% CI 2-sided [-32.7 to -11.5] — Response Rate Difference = Upadacitinib - Placebo

34. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 12 Points From Baseline in ADerm-IS Sleep Domain Score at Week 16
Description: The ADerm-IS is a 10-item patient reported outcome questionnaire designed to assess a variety of impacts that participants experience from their AD.
  The ADerm-IS sleep domain consists of 3 questions designed to assess the impact of AD on sleep on a daily basis over a 24-hour recall period. The items include difficulty falling asleep, impact on sleep, and waking at night. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The ADerm-IS sleep domain score is the sum of the 3 item scores and ranges from 0 (no impact) to 30 (worst impact). The ADerm-IS sleep domain was analyzed based on weekly rolling averages of daily scores.
  The minimal clinically important difference for ADerm-IS sleep domain score is 12.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with ADerm-IS Sleep Domain score ≥ 12 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 48 | 49 | 47
percentage of participants | 12.5 [3.1 to 21.9] | 46.9 [33.0 to 60.9] | 66.0 [52.4 to 79.5]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 53.6, 95% CI 2-sided [37.7 to 69.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 34.8, 95% CI 2-sided [18.1 to 51.4] — Response Rate Difference = Upadacitinib - Placebo

35. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in ADerm-SS Skin Pain Score at Week 16
Description: The ADerm-SS is an 11-item PRO questionnaire designed to assess signs and symptoms that patients may experience due to AD using a 24-hour recall period. For the skin pain item participants were asked to indicate on a daily basis how bad their worst skin pain due to AD was in the past 24 hours on an NRS from 0 (no pain) to 10 (worst imaginable pain). The minimal clinically important difference for ADerm-SS skin pain score is 4.
  The ADerm-SS skin pain score was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with ADerm-SS Skin Pain score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 44 | 54 | 59
percentage of participants | 9.1 [0.6 to 17.6] | 42.6 [29.4 to 55.8] | 64.4 [52.2 to 76.6]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 56.6, 95% CI 2-sided [42.0 to 71.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 32.5, 95% CI 2-sided [16.9 to 48.1] — Response Rate Difference = Upadacitinib - Placebo

36. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 28 Points From Baseline in ADerm-SS TSS-7 at Week 16
Description: as for outcome 13
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with ADerm-SS TSS-7 ≥ 28 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 49 | 52 | 55
percentage of participants | 16.3 [6.0 to 26.7] | 51.9 [38.3 to 65.5] | 67.3 [54.9 to 79.7]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 50.9, 95% CI 2-sided [35.1 to 66.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 35.7, 95% CI 2-sided [18.8 to 52.6] — Response Rate Difference = Upadacitinib - Placebo

37. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 11 Points From Baseline in ADerm-IS Emotional State Domain Score at Week 16
Description: as for outcome 14
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with ADerm-IS Emotional State Domain score ≥ 11 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 46 | 47 | 47
percentage of participants | 23.9 [11.6 to 36.2] | 61.7 [47.8 to 75.6] | 78.7 [67.0 to 90.4]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 54.4, 95% CI 2-sided [37.4 to 71.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 38.1, 95% CI 2-sided [19.8 to 56.4] — Response Rate Difference = Upadacitinib - Placebo

38. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 14 Points From Baseline in ADerm-IS Daily Activities Domain Score at Week 16
Description: as for outcome 15
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with ADerm-IS Daily Activities Domain Score ≥ 14 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 43 | 43 | 43
percentage of participants | 30.2 [16.5 to 44.0] | 58.1 [43.4 to 72.9] | 81.4 [69.8 to 93.0]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 51.2, 95% CI 2-sided [33.3 to 69.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 28.1, 95% CI 2-sided [8.0 to 48.2] — Response Rate Difference = Upadacitinib - Placebo

39. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 100 Response at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 100 response is defined as a 100% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 16
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 61 | 64 | 64
percentage of participants | 0.0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 15.6 [6.7 to 24.5] | 31.3 [19.9 to 42.6]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 31.2, 95% CI 2-sided [19.9 to 42.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 15.8, 95% CI 2-sided [6.9 to 24.6] — Response Rate Difference = Upadacitinib - Placebo

40. Secondary Outcome: Adolescents: Percent Change From Baseline in Worst Pruritus NRS at Week 16
Description: as for outcome 17
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with non-missing Baseline and Week 16 values; missing data were handled using a mixed-effect model with repeated measurements including observed measurements at all visits, except that measurements after any rescue medication were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 34 | 50 | 57
percent change | -24.40 [-35.03 to -13.78] | -58.28 [-67.23 to -49.33] | -66.82 [-75.57 to -58.07]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, and Baseline vIGA-AD category in the model; LS Mean Difference = -42.42, 95% CI 2-sided [-56.16 to -28.68] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 40, analysis 1]; LS Mean Difference = -33.88, 95% CI 2-sided [-47.76 to -19.99] — Difference = Upadacitinib - Placebo

41. Secondary Outcome: Adolescents: Percent Change From Baseline in EASI Score at Week 16
Description: as for outcome 18
Time Frame: Baseline and Week 16
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 33 | 60 | 63
percent change | -43.19 [-51.15 to -35.24] | -81.04 [-87.67 to -74.41] | -85.03 [-91.56 to -78.50]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 40, analysis 1]; LS Mean Difference = -41.84, 95% CI 2-sided [-52.09 to -31.58] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 40, analysis 1]; LS Mean Difference = -37.84, 95% CI 2-sided [-48.17 to -27.52] — Difference = Upadacitinib - Placebo

42. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in POEM Total Score at Week 16
Description: as for outcome 19
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with POEM score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 58 | 63 | 64
percentage of participants | 31.0 [19.1 to 42.9] | 81.0 [71.3 to 90.6] | 85.9 [77.4 to 94.5]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 54.8, 95% CI 2-sided [40.3 to 69.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 50.0, 95% CI 2-sided [34.8 to 65.3] — Response Rate Difference = Upadacitinib - Placebo

43. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in DLQI Score at Week 16
Description: as for outcome 20
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents who were ≥ 16 years old at Screening with DLQI score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 22 | 28 | 32
percentage of participants | 36.4 [16.3 to 56.5] | 82.1 [68.0 to 96.3] | 81.3 [67.7 to 94.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 45.1, 95% CI 2-sided [21.0 to 69.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 49.6, 95% CI 2-sided [26.7 to 72.5] — Response Rate Difference = Upadacitinib - Placebo

44. Secondary Outcome: Adolescents: Percent Change From Baseline in SCORAD Score at Week 16
Description: as for outcome 21
Time Frame: Baseline and Week 16
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 33 | 59 | 63
percent change | -32.52 [-40.95 to -24.08] | -65.22 [-71.87 to -58.56] | -71.44 [-77.91 to -64.97]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, and Baseline vIGA-AD category; LS Mean Difference = -38.92, 95% CI 2-sided [-49.54 to -28.31] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 44, analysis 1]; LS Mean Difference = -32.70, 95% CI 2-sided [-43.44 to -21.96] — Difference = Upadacitinib - Placebo

45. Secondary Outcome: Adolescents: Percentage of Participants Achieving HADS-A Score and HADS-D Score of < 8 at Week 16
Description: as for outcome 22
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with HADS-A ≥ 8 or HADS-D ≥ 8 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 26 | 35 | 27
percentage of participants | 3.8 [0.0 to 11.2] | 48.6 [32.0 to 65.1] | 55.6 [36.8 to 74.3]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 51.7, 95% CI 2-sided [31.7 to 71.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 44.7, 95% CI 2-sided [26.7 to 62.8] — Response Rate Difference = Upadacitinib - Placebo

46. Secondary Outcome: Adolescents: Percentage of Participants Achieving a DLQI Score of 0 or 1 at Week 16
Description: as for outcome 23
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents who were ≥ 16 years old at Screening with DLQI score ≥ 1 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 22 | 28 | 33
percentage of participants | 4.5 [0.0 to 13.2] | 21.4 [6.2 to 36.6] | 30.3 [14.6 to 46.0]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 25.1, 95% CI 2-sided [7.3 to 43.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.093, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 15.8, 95% CI 2-sided [-2.6 to 34.2] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 16, or 30 days after last dose for participants who did not enter the blinded extension period.
Groups:
- Adults: Upadacitinib 15 mg QD: Participants ≥ 18 years old received upadacitinib 15 mg orally once daily for 16 weeks.
- Adults: Upadacitinib 30 mg QD: Participants ≥ 18 years old received upadacitinib 30 mg orally once daily for 16 weeks.
- Adolescents: Placebo: Adolescent participants (12 - 17 years old) received placebo orally once a day (QD) for 16 weeks.
- Adolescents: Upadacitinib 15 mg QD: Adolescent participants (12 - 17 years old) received upadacitinib 15 mg orally once daily for 16 weeks.
- Adolescents: Upadacitinib 30 mg QD: Adolescent participants (12 - 17 years old) received upadacitinib 30 mg orally once daily for 16 weeks.
Arm/Group | Adults: Placebo | Adults: Upadacitinib 15 mg QD | Adults: Upadacitinib 30 mg QD | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/239 | 0/243 | 0/61 | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 7/241 | 5/239 | 8/243 | 1/61 | 1/64 | 0/64
Other Adverse Events (participants affected / at risk) | 64/241 | 67/239 | 102/243 | 13/61 | 19/64 | 25/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults: Placebo (N=241) | Adults: Upadacitinib 15 mg QD (N=239) | Adults: Upadacitinib 30 mg QD (N=243) | Adolescents: Placebo (N=61) | Adolescents: Upadacitinib 15 mg QD (N=64) | Adolescents: Upadacitinib 30 mg QD (N=64)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOD ALLERGY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMPETIGO (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults: Placebo (N=241) | Adults: Upadacitinib 15 mg QD (N=239) | Adults: Upadacitinib 30 mg QD (N=243) | Adolescents: Placebo (N=61) | Adolescents: Upadacitinib 15 mg QD (N=64) | Adolescents: Upadacitinib 30 mg QD (N=64)
NASOPHARYNGITIS (Infections and infestations) | 15 (17) | 19 (19) | 28 (35) | 1 (1) | 3 (3) | 5 (5)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 (19) | 20 (21) | 31 (35) | 5 (6) | 5 (6) | 8 (9)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 5 (5) | 12 (14) | 11 (13) | 2 (2) | 5 (6) | 5 (5)
HEADACHE (Nervous system disorders) | 10 (12) | 12 (13) | 16 (16) | 2 (2) | 5 (6) | 4 (5)
ACNE (Skin and subcutaneous tissue disorders) | 6 (6) | 13 (14) | 40 (42) | 1 (1) | 8 (8) | 10 (10)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 22 (23) | 8 (8) | 4 (4) | 2 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT03569293/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03569293/SAP_001.pdf